CLINICAL TRIAL: NCT02635373
Title: European Calciphylaxis Registry Network
Acronym: EuCalNet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 13-093
Record Dates: First submitted 2015-11-25; First posted 2015-12-18 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Calcific Uremic Arteriolopathy (CUA); Calciphylaxis
Keywords: Calciphylaxis; Rare disease (ORPHA280062); Renal insufficiency; ESRD; Calcification; Chronic kidney disease; Dialysis; Vascular disease
MeSH Terms: conditions — Calciphylaxis; Rare Diseases; Renal Insufficiency; Kidney Failure, Chronic; Calcinosis; Renal Insufficiency, Chronic; Vascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational, registry, prospective, non-interventional collection of CUA patient data. Patient treatment is carried out within clinical routine, at the discretion of the physicians and according to existing treatment guidelines. Participating physicians will not be subject to any instructions with regard to the diagnosis and therapy of their patients.

DETAILED DESCRIPTION:
Calcific uremic arteriolopathy (CUA, calciphylaxis) is a rare disease (ORPHA280062) with dramatically high mortality characterized clinically by the occurrence of painful debilitating cutaneous lesions and ulcerations. Median survival time is about 1.5 years. Many uncertainties still exist about risk factors and optimal therapy. CUA mainly occurs in patients with severe renal insufficiency or ESRD.

The aim of the present initiative is to establish an international (European) observational registry for CUA patients. This registry will help to reach a critical mass of CUA patients, will allow novel insights into pathophysiology, and will help establishing systematically an overview upon risk factors and long-term outcome of CUA patients. The design of the international registry is supposed to adopt the structure of the presently running nation-wide German calciphylaxis registry.

The investigators plan to initiate a registry in which treating physicians can provide data upon demographics, clinical picture, comorbidities, medical treatments and laboratory data at the time of diagnosis and serial follow-up time points. In addition investigators will build-up a biobank for full blood, serum and plasma samples as well as tissue samples.

The registry will allow investigations regarding potential subgroups of patients (proximal versus distal forms of CUA), geno-phenotype correlations, description of international state-of-the-art treatment, and identification of preventive tools, risk factors and biomarkers for estimation of prognosis.

Furthermore, the registry will be the nidus for further scientific exchange between experts and clinicians on the field of uremic vascular calcification.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed CUA according to the judgement of locally treating physicians, who have the option to ask for external diagnostic advice from the country-specific sub-investigators
* Male or female aged > 18 years
* Written informed consent prior to study participation
* The subject is not mentally or legally incapacitated

Exclusion Criteria:

• The subject is not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed CUA
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Prognosis of patients with calciphylaxis (survival time) | 5 years
  Survival time is defined as 1) time between diagnosis of calciphylaxis and death (or end of follow-up) or 2) - in case time of diagnosis is not recorded - time between registry recording and death (or end of follow-up). Analysis of survival time is done using the Kaplan-Meier survival analysis and Kaplan-Meier plot. With a Cox hazard model, we will try to identify additional factors influencing survival time. Hereby it is possible to take into consideration interaction between the parameters.

SECONDARY OUTCOMES:
Diagnosis of calciphylaxis | 5 years
  An internet based multilingual registry in which treating physicians can provide patients' data (online questionnaire) upon: demographics, the clinical picture including photo documentation and pain scale (VAS) reporting, comorbidities, medical treatments including dialysis and operations, wound management and laboratory data (serum-creatinine, , BUN, ionized / total calcium, serum phosphorus, PTH, alkaline, phosphatase, calcidiol, albumin, CRP, HbA1c, cholesterol, ferritin, hemoglobin, leukocyte count). The international registry will allow a more rapid identification of patients with calciphylaxis than on a national basis alone, will help establish diagnostic algorithms, and will increase the awareness of the disease.
Risk factors | 5 years
  More detailed identification of risk factors: the registry will allow investigations regarding potential subgroups of patients (proximal versus distal forms of CUA), geno-phenotype correlations, description of international state-of-the-art treatment, and identification of preventive tools, risk factors and biomarkers for estimation of prognosis.
Factors influencing prognosis of patients with calciphylaxis | 5 years
  Evaluation of the collected data from the time point of diagnosis and serial follow-up time points and further scientific exchange between experts and clinicians on the field of uremic vascular calcification will allow identification of subgroups of patients with potentially distinct pattern of risk factors, clinical picture and prognosis, and establishing factors influencing prognosis of patients with calciphylaxis and to develop novel and/or individualized treatment strategies
Novel therapeutic options | 5 years
  By increasing the reported cases towards a critical threshold in Europe enabling the performance of RCTs comparing available or upcoming therapeutic options in CUA pts.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonary Diseases and Vascular Medicine at the University Hospital, RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Weenig RH. Pathogenesis of calciphylaxis: Hans Selye to nuclear factor kappa-B. J Am Acad Dermatol. 2008 Mar;58(3):458-71. doi: 10.1016/j.jaad.2007.12.006. Epub 2008 Jan 18. PMID 18206262
- [Background] Brandenburg VM, Cozzolino M, Ketteler M. Calciphylaxis: a still unmet challenge. J Nephrol. 2011 Mar-Apr;24(2):142-8. doi: 10.5301/jn.2011.6366. PMID 21337312
- [Background] Meissner M, Gille J, Kaufmann R. Calciphylaxis: no therapeutic concepts for a poorly understood syndrome? J Dtsch Dermatol Ges. 2006 Dec;4(12):1037-44. doi: 10.1111/j.1610-0387.2006.06127.x. English, German. PMID 17176411
- [Background] Hafner J, Keusch G, Wahl C, Sauter B, Hurlimann A, von Weizsacker F, Krayenbuhl M, Biedermann K, Brunner U, Helfenstein U. Uremic small-artery disease with medial calcification and intimal hyperplasia (so-called calciphylaxis): a complication of chronic renal failure and benefit from parathyroidectomy. J Am Acad Dermatol. 1995 Dec;33(6):954-62. doi: 10.1016/0190-9622(95)90286-4. PMID 7490365
- [Background] Mazhar AR, Johnson RJ, Gillen D, Stivelman JC, Ryan MJ, Davis CL, Stehman-Breen CO. Risk factors and mortality associated with calciphylaxis in end-stage renal disease. Kidney Int. 2001 Jul;60(1):324-32. doi: 10.1046/j.1523-1755.2001.00803.x. PMID 11422768
- [Background] Janigan DT, Hirsch DJ, Klassen GA, MacDonald AS. Calcified subcutaneous arterioles with infarcts of the subcutis and skin ("calciphylaxis") in chronic renal failure. Am J Kidney Dis. 2000 Apr;35(4):588-97. doi: 10.1016/s0272-6386(00)70003-5. PMID 10739777
- [Background] Kramann R, Brandenburg VM, Schurgers LJ, Ketteler M, Westphal S, Leisten I, Bovi M, Jahnen-Dechent W, Knuchel R, Floege J, Schneider RK. Novel insights into osteogenesis and matrix remodelling associated with calcific uraemic arteriolopathy. Nephrol Dial Transplant. 2013 Apr;28(4):856-68. doi: 10.1093/ndt/gfs466. Epub 2012 Dec 6. PMID 23223222
- [Background] Fine A, Zacharias J. Calciphylaxis is usually non-ulcerating: risk factors, outcome and therapy. Kidney Int. 2002 Jun;61(6):2210-7. doi: 10.1046/j.1523-1755.2002.00375.x. PMID 12028462
- [Background] Weenig RH, Sewell LD, Davis MD, McCarthy JT, Pittelkow MR. Calciphylaxis: natural history, risk factor analysis, and outcome. J Am Acad Dermatol. 2007 Apr;56(4):569-79. doi: 10.1016/j.jaad.2006.08.065. Epub 2006 Dec 1. PMID 17141359
- [Background] Brandenburg VM, Floege J, Ketteler M. Kalzifizierende urämische Arteriolopathie. Der Nephrologe 2009; 4(1):65-66
- [Background] Krueger T, Westenfeld R, Schurgers L, Brandenburg V. Coagulation meets calcification: the vitamin K system. Int J Artif Organs. 2009 Feb;32(2):67-74. doi: 10.1177/039139880903200202. PMID 19363777
- [Background] Jahnen-Dechent W, Schafer C, Ketteler M, McKee MD. Mineral chaperones: a role for fetuin-A and osteopontin in the inhibition and regression of pathologic calcification. J Mol Med (Berl). 2008 Apr;86(4):379-89. doi: 10.1007/s00109-007-0294-y. Epub 2007 Dec 15. PMID 18080808
- [Background] Cranenburg EC, Vermeer C, Koos R, Boumans ML, Hackeng TM, Bouwman FG, Kwaijtaal M, Brandenburg VM, Ketteler M, Schurgers LJ. The circulating inactive form of matrix Gla Protein (ucMGP) as a biomarker for cardiovascular calcification. J Vasc Res. 2008;45(5):427-36. doi: 10.1159/000124863. Epub 2008 Apr 10. PMID 18401181
- [Background] Schafer C, Heiss A, Schwarz A, Westenfeld R, Ketteler M, Floege J, Muller-Esterl W, Schinke T, Jahnen-Dechent W. The serum protein alpha 2-Heremans-Schmid glycoprotein/fetuin-A is a systemically acting inhibitor of ectopic calcification. J Clin Invest. 2003 Aug;112(3):357-66. doi: 10.1172/JCI17202. PMID 12897203